CLINICAL TRIAL: NCT06070870
Title: Health Education Approach to Lung Screening (HEALS)
Brief Title: Health Education Approach to Lung Screening
Acronym: HEALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SU2C-WINN; HM20026222 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Screening
MeSH Terms: conditions — Lung Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Navigation (Experimental): Centralized patient navigators will be trained to help patients navigate the clinical, logistical, and financial aspects of LCS. Navigators employ case management approaches based on social work principles. The experience of patient navigation will be tailored to the individual participant
  Interventions: Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: Patient Navigation — Navigation will address the following 4 domains of barriers to screening:
  * Individual
  * Organizational
  * Economic
  * Sociocultural At the first visit, navigators will assess the participant's barriers in each of these domains. Any follow-up visits, if necessary, will be used to help the participant overcome these barriers to screening

SUMMARY:
Evaluate the impact of the patient navigation program on the proportion of patients who complete lung cancer screening (LCS), defined as undergoing a low dose computed tomography (LDCT)

DETAILED DESCRIPTION:
This is a single-arm study of a patient navigation intervention to increase access to lung cancer screening (LCS).

ELIGIBILITY:
Inclusion Criteria:

* Meets current USPSTF guidelines for lung cancer screening (LCS)
* 20 pack-year smoking history Note: A pack-year is a way of calculating how much a person has smoked in their lifetime.

One pack-year is the equivalent of smoking an average of 20 cigarettes-1 pack-per day for a year.

* Currently smokes or has quit smoking within the past 15 years
* Identifies as Black or African-American Note: Both Hispanic/Latino and Non-Hispanic/Latino patients are eligible as long as they also identify as Black or African-American (eg, Afro-Latino).
* Willing to complete all navigation-related study activities
* Able to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

A patient who meets any of the following exclusion criteria is ineligible to participate in the study:

* Known history of cancer (except squamous cell skin cancer), or coughing up blood in the past 5 years, as reported by the individual
* Has undergone a previous lung cancer screening
* Inability to speak English
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of study patients who complete lung cancer screening (LCS) through the patient navigation process | 2 weeks to 4 months following day 1, varies by participant
  Evaluate the impact of the patient navigation program on the number of patients who complete lung cancer screening (LCS), defined as undergoing a low dose computed tomography (LDCT).

SECONDARY OUTCOMES:
Assess the feasibility and acceptability of the patient navigation program | Day 1
  Determine the number of participants that are satisfied with the navigation program by utilizing Was It Worth It instrument; that consists of 8 items that are are answered "yes", "no" or "uncertain".
Assess the feasibility and acceptability of the patient navigation program | 2 weeks to 4 months following day 1, varies by participant
  Determine the number of participants that are satisfied with the navigation program by utilizing Was It Worth It instrument; that consists of 8 items that are are answered "yes", "no" or "uncertain" after the navigation program.
Assess the impact of the patient navigation program on patient health-related quality of life at baseline. | Day 1
  Utilizing Patient-Reported Outcome Measurement Information System (PROMIS) v1.2 Global Health Scale (10 items) scores before and after navigation intervention. Patient-Reported Outcome Measurement Information System (PROMIS) v1.2 Global Health Scale (10 items), measures assess physical, mental, and social health where 5=Never, 4=Rarely, 3=Sometimes, 2=Often, and 1=Always. Higher scores indicate better health.
Assess the impact of the patient navigation program on patient health-related quality of life after navigation intervention. | 2 weeks to 4 months following day 1, varies by participant
  Utilizing Patient-Reported Outcome Measurement Information System (PROMIS) v1.2 Global Health Scale (10 items) scores before and after navigation intervention. Patient-Reported Outcome Measurement Information System (PROMIS) v1.2 Global Health Scale (10 items), measures assess physical, mental, and social health, where 5=Never, 4=Rarely, 3=Sometimes, 2=Often, and 1=Always. Higher scores indicate better health.
Assess the impact of the patient navigation program on patient financial distress | Day 1
  Determine the number of participants that have financial distress at baseline utilizing Financial Distress measure scores at baseline. Study-specific financial distress measure (8 items) each item will need to be individually coded 1-5, with 1=completely disagree to 5=completely agree and 98 for Don't know and 99 for Not applicable.
Assess the impact of the patient navigation program on patient financial distress | 2 weeks to 4 months following day 1, varies by participant
  Determine the number of participants that have lessening financial distress after the navigation program utilizing Financial Distress measure scores at baseline. Study-specific financial distress measure (8 items) each item will be individually coded 1-5, with 1=completely disagree to 5=completely agree and 98 for Don't know and 99 for Not applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Sheppard, PhD, Principal Investigator — Virginia Commonwealth University
Locations (3):
- United States (3):
  - University of North Carolina-Chapel Hill, Carrboro, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
Currently there is not a plan to share with other researchers not working on the protocol.